CLINICAL TRIAL: NCT04033627
Title: A Multi-center Prospective Clinical Study in China Using CliniMACS TCRα/β+ and CD45RA+ T Cell Depleted Stem Cell Grafts From Haploidentical Donors for Hematopoietic Stem Cell Transplantation in Children With Leukemia
Brief Title: TCDαβ/CD45RA Haploidentical Transplantation in Children With Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Children's Hospital of Soochow University (Other); Chinese University of Hong Kong (Other); Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD Haplo
Record Dates: First submitted 2019-06-12; First posted 2019-07-26 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Relapsed Pediatric ALL; Acute Graft-Versus-Host Disease (Gvhd) Grade IV (Diagnosis); Relapsed Pediatric AML
Keywords: In Vitro T cell depletion; haploidentical transplantation; GVHD; leukemia; TCRab; CD45RA; CliniMACS
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Graft vs Host Disease; Disease; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In Vitro T cell depletion (Experimental): Use the CliniMACS TCRα/β and CD45 Systems to deplete TCRα/β+ and CD45RA+ cells from the mobilized peripheral blood stem cells of a haploidentical donor in patients with leukemia.
  Interventions: Procedure: In Vitro T cells depletion using CliniMCAS system

INTERVENTIONS:
Procedure: In Vitro T cells depletion using CliniMCAS system — Use the CliniMACS TCRα/β and CD45 Systems to deplete TCRα/β+ and CD45RA+ cells from the mobilized peripheral blood stem cells of a haploidentical donor in patients with leukemia.

SUMMARY:
This is a multi-center clinical study in China using CliniMACS TCRα/β+ and CD45RA+ T cell depleted stem cell grafts from haploidentical donors for hematopoietic stem cell transplantation in children.

DETAILED DESCRIPTION:
This clinical study will the CliniMACS TCRα/β and CD45RA Systems to deplete TCRα/β+ and CD45RA+ cells from the mobilized peripheral blood stem cells of a haploidentical donors to treat pediatric patients who were suffuring form relapsed or refactory leukemia.

Aming to evaluate the safety/tolerability and feasibility of haploidentical PBSC grafts depleted of TCRα/β+ and CD45RA+ cells using the CliniMACS TCRαβ/CD45RA System in pediatric patients with hematological malignancies diseases. And the incidence of grade II-IV acute graft-versus-host disease (GVHD) until Day 100 post-transplantation of this new In Vitro T cell depletion technology in China.

The investigators will monitor the incidence of grade I acute GVHD until Day 100 post-transplantation, incidence and severity of chronic GVHD after 1 year and 2 years, incidence of NRM at all visits throughout the study, and graft failure from Day 0 to Day 28 at the same time.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients with hematological malignancies in complete remission (CR), partial remission (PR) or with stable disease

* Acute myeloid leukemia (AML):

Patients with high-risk AML in CR1 Patients with relapsed or primary therapy-refractory AML

* Acute lymphoid leukemia (ALL):

Patients with high-risk ALL in CR1 Patients with relapsed or primary refractory ALL

Exclusion Criteria:

* Age >18 years or <8 weeks
* Patients with progressive disease prior HCT
* <3 months after preceding hematopoietic cell transplantation (HCT)
* History of neurological impairment (active seizures, severe peripheral neuropathy, signs of leukencephalopathy, active CNS infection)
* Fungal infections with radiological and clinical progression
* Liver function abnormalities with bilirubin >2 mg/dL and elevation of transaminases higher than 400 U/L
* Chronic active viral hepatitis
* Ejection fraction <40% or shortening fraction <25% on echocardiography
* Patients with > grade II hypertension by Common Toxicity Criteria (CTC)
* Creatinine clearance below threshold defined for stem cell transplantation according to local clinical standard
* Respiratory failure necessitating supplemental oxygen
* HIV infection
* Concurrent severe or uncontrolled medical disease (e.g. uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months prior to the study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) which by assessment of the treating physician could compromise participation in the study
* Patients with a history of psychiatric illness or a condition which could interfere with their ability to understand the requirements of the study (this includes alcoholism/drug addiction)
* Patients unwilling or unable to comply with the protocol or unable to give informed consent
* Treatment with any investigational product within 4 weeks prior to study treatment (transfusion of the IMP)

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2024-05-08 (Estimated)

PRIMARY OUTCOMES:
Log number of In Vitro T cells depletion | One week
  Log number of In Vitro T cells depletion using CliniMACS TCRab/CD45RA system.
Incidence of grade II-IV acute GVHD | up to 3 months
  Incidence of grade II-IV acute graft-versus-host disease (GVHD) until Day 100 post-transplantation.

SECONDARY OUTCOMES:
Grade I aGVHD | up to 3 months
  Incidence of grade I acute GVHD until Day 100 post-transplantation
cGVHD | 2 years
  Incidence and severity of chronic GVHD in 1 year and 2 years
NRM | 1 year
  Incidence of NRM at all visits throughout the study
Graft failure | 1 month
  incidence of Graft failure from Day 0 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No